CLINICAL TRIAL: NCT05616871
Title: Real-world Effectiveness and Treatment Patterns of Upadacitinib in Monotherapy or Used in Combination With Methotrexate in Active Psoriatic Arthritis Patients
Brief Title: An Observational Study to Assess Change in Disease Activity and Treatment Patterns of Upadacitinib When Given Alone or Co-Administered With Methotrexate in Adult Participants With Active Psoriatic Arthritis
Acronym: UPtimum-PsA
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P22-897
Record Dates: First submitted 2022-11-09; First posted 2022-11-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA; UPA; Upadacitinib; Rinvoq®
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib Alone or In Combination with Methotrexate: Participants will receive upadacitinib alone or in combination with methotrexate as prescribed by their physician according to local label in real- world practice.

SUMMARY:
Psoriatic arthritis (PsA) is a chronic, immune-mediated, systemic disease affecting less than 1% of people with variations by parts of the world, and around 20%-30% of participants with psoriasis.

Upadacitinib (RINVOQ) is approved drug for the treatment of adult participants with active PsA in Europe. Approximately 450 adult participants who are prescribed Upadacitinib by their physician in accordance with local label will be enrolled in 4 countries in Europe: France, Germany, Greece and Italy.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 24 months.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of active psoriatic arthritis (PsA) whose peripheral involvement justifies the prescription of upadacitinib upon judgement of the treating physician.
* Physician decision on participant treatment with upadacitinib must have been reached prior to and independently of recruitment in the study.
* Upadacitinib prescribed in accordance with the applicable approved label and local regulatory and reimbursement policies.
* Participants able to understand and communicate with the investigator and comply with the requirements of the study.

Exclusion Criteria:

* Participation in a clinical trial of an investigational drug, concurrently or within the last 30 days.
* Prior treatment with upadacitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with Psoriatic Arthritis (PsA)
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Disease Activity in Psoriatic Arthritis (DAPSA): score <=14 | Month 6
  Disease Activity in Psoriatic Arthritis (DAPSA) score is calculated by the sum of values of rheumatic parameters [tender joint count (TJC/ 68) + swollen joint count (SJC/ 66) + visual analog scale VAS Patient Global Disease Activity (PtGA) in cm + VAS Patient Pain in cm + C Reactive Protein (CRP) in mg/dL].

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (88):
- France (37):
  - Centre Hospitalier Universitaire de Nice - Hôpital Pasteur /ID# 252536, Nice, Alpes-Maritimes
  - CH Troyes - Hopital Simone Veil /ID# 252625, Troyes, Aube
  - CHU de Besancon - Jean Minjoz /ID# 252537, Besançon, Doubs
  - CHU Limoges - Dupuytren 1 /ID# 252432, Limoges, Franche-Comte
  - CHU Toulouse - Hopital Purpan /ID# 252077, Toulouse, Haute-Garonne
  - CHU Montpellier - Hopital Saint Eloi /ID# 252078, Montpellier, Herault
  - CHU Grenoble - Hopital Michallon /ID# 252601, La Tronche, Isere
  - CHU Bordeaux - Hopital Pellegrin /ID# 252532, Bordeaux, Nouvelle-Aquitaine
  - Ch Beauvais /Id# 252464, Beauvais, Oise
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 245194, Créteil, Paris
  - Infirmerie Protestante /ID# 252075, Caluire-et-Cuire, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 252527, Amiens, Somme
  - Cabinet libéral du Dr PAUPIERE /ID# 252604, Péronne, Somme
  - Chic Castres-Mazamet /Id# 259557, Castres, Tarn
  - CH Henri Duffaut /ID# 252620, Avignon, Vaucluse
  - CHD Vendée- La Roche-sur-Yon - Les Oudairies /ID# 259549, La Roche-sur-Yon, Vendee
  - CH AIX LES BAIN - Reine Hortense /ID# 252465, Aix-les-Bains
  - Cabinet Médical Dr ALBERT-SABONNADIERE /ID# 252523, Antibes
  - Centre Hospitalier d'Arras /ID# 252529, Arras
  - Centre Hospitalier de Boulogne Sur Mer /ID# 252467, Boulogne-sur-Mer
  - Centre Hospitalier Jean Rougie /ID# 259550, Cahors
  - CH de Cannes - Simone Veil /ID# 252600, Cannes
  - CHRU Tours - Hopital Trousseau /ID# 252528, Chambray-lès-Tours
  - C. H. Sud Francilien /ID# 254945, Corbeil-Essonnes
  - CH La Rochelle - Hopital Saint Louis /ID# 252534, La Rochelle
  - Hopital St Joseph - St Luc (Lyon) /ID# 259561, Lyon
  - Clinique de la Sauvegarde /ID# 252533, Lyon
  - ELSAN - Clinique du Pont de Chaume /ID# 252602, Montauban
  - CH de Narbonne /ID# 252525, Narbonne
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 252530, Orléans
  - AP-HP - Groupe Hospitalier 10e - Hopital Lariboisiere /ID# 252526, Paris
  - AP-HP - Hopital Saint-Antoine /ID# 252627, Paris
  - AP-HP - Hopital Bichat - Claude-Bernard /ID# 252531, Paris
  - GH Diaconesses Croix Saint-Simon /ID# 252463, Paris
  - CHU de Rennes - Hospital Sud /ID# 252478, Rennes
  - Hôpital Charles-Nicolle /ID# 252603, Rouen
  - Cabinet Du Dr Judith Payet Dubourg /Id# 252668, Saint-Pierre-des-Corps
- Germany (19):
  - Rheumazentrum Ruhrgebiet /ID# 252939, Herne, North Rhine-Westphalia
  - Beyer, Kaiserslautern, DE /ID# 254754, Kaiserslautern, Rhineland-Palatinate
  - Krankenhaus der Barmherzigen Brüder Trier /ID# 254762, Trier, Rhineland-Palatinate
  - Dr. Murawski /ID# 257911, Neunkirchen, Saarland
  - Rheumapraxis Dr. Prothmann /ID# 254759, Püttlingen, Saarland
  - Aurich & Sieburg, Magdeburg /ID# 255504, Magdeburg, Saxony-Anhalt
  - MVZ Ambulantes Rheumazentrum Erfurt /ID# 256115, Erfurt, Thuringia
  - Kupka & Kupka, Altenburg, DE /ID# 254758, Altenburg
  - Rheumatologische Schwerpunktpraxis Brandt-Juergens /ID# 258152, Berlin
  - Praxis Dr. Silke Zinke /ID# 258037, Berlin
  - MVZ Herzogin Elisabeth Hospital /ID# 266740, Braunschweig
  - Praxis Dilltal /ID# 254761, Ehringshausen
  - Universitaetsmedizin Greifswald /ID# 254756, Greifswald
  - Dr. Heintz /ID# 254757, Hamburg
  - Dr. Bolze, Ludwigshafen, DE /ID# 254134, Ludwigshafen
  - RHIO Forschungsinstitut /ID# 254752, Meerbusch
  - Prof-med-stud.de /ID# 265965, Munich
  - Knappschaftsklinikum Saar /ID# 255505, Püttlingen
  - Krankenhaus St. Josef /ID# 254755, Wuppertal
- Greece (20):
  - Olympion General Clinic /ID# 247644, Pátrai, Achaia
  - 251 Airforce General Hospital /ID# 248092, Athens, Attica
  - Henry Dunnant Hospital Center /ID# 247640, Athens, Attica
  - General Hospital of Athens Gennimatas /ID# 247635, Athens, Attica
  - General Hospital of Athens Ippokratio /ID# 247633, Athens, Attica
  - General Hospital of Athens Laiko /ID# 247634, Athens, Attica
  - General Hospital of Athens Laiko /ID# 258030, Athens, Attica
  - University General Hospital Attikon /ID# 248093, Athens, Attica
  - General Hospital of Elefsina Thriassio /ID# 251900, Magoula (Attikis), Attica
  - Iaso /ID# 247649, Marousi, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 247632, Heraklion, Crete
  - Naval Hospital of Athens /ID# 247631, Athens
  - KAT Atttica General Hospital /ID# 247641, Athens
  - University General Hospital of Ioannina /ID# 251899, Ioannina
  - Iaso Thessalias S.A. /Id# 255110, Larissa
  - Reg Gen Univ Hosp Larissa /ID# 247642, Larissa
  - Bioclinic Thessaloniki /ID# 247648, Thessaloniki
  - Euromedica Blue Cross Gen Clin /ID# 251898, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 247643, Thessaloniki
  - Euromedica General Clinic /ID# 251897, Thessaloniki
- Italy (12):
  - IRCCS Istituto Clinico Humanitas /ID# 251275, Rozzano, Lombardy
  - IRCCS Ospedale San Raffaele /ID# 251562, Milan, Milano
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 251183, Naples, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 250817, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 250669, Rome, Roma
  - Azienda Ospedaliero Universitaria delle Marche /ID# 250819, Ancona
  - A.O.U. Consorziale Policlinico di Bari /ID# 251508, Bari
  - Universita degli Studi del Molise /ID# 251176, Campobasso
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone /ID# 250789, Palermo
  - Fondazione IRCCS Policlinico San Matteo /ID# 250747, Pavia
  - Azienda Ospedaliera Universitaria Senese /ID# 251146, Siena
  - Azienda Ospedaliera Universitaria Friuli Centrale/Presidio Ospedaliero Universit /ID# 251544, Udine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.rxabbvie.com/